CLINICAL TRIAL: NCT00150826
Title: A Double-Blind, Multicenter, Placebo Controlled Study of Quinapril in Women With Chest Pain, Coronary Flow Reserve Limitations and Evidence of Myocardial Ischemia in the Absence of Significant Epicardial Coronary Artery Disease.
Brief Title: QWISE - Study of Quinapril in Women With Chest Pain, Coronary Flow Reserve Limitations and Evidence of Myocardial Ischemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QWISE; 5U01HL064924-04 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Ischemic Heart Disease
Keywords: microvascular disease; women; renin angiotensin system; WISE; ischemic heart disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Quinapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quinapril (Active Comparator): This arm will receive quinapril which will be started at 40mg daily and titrated to 80mg daily by the end of the first week. After treatment on the maximum tolerated dose for 16 weeks, patients will be reevaluated with coronary angiogram with coronary flow reserve measurements and assessment of angina using the Seattle Angina Questionnaire.
  Interventions: Drug: Quinapril
- Placebo (Placebo Comparator): This arm will receive placebo for 16 weeks and will be reevaluated with coronary angiogram with coronary flow reserve measurements and assessment of angina using the Seattle Angina Questionnaire.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinapril — Quinapril will be started at 40mg daily and titrated to 80mg daily for 16 weeks.
  Arms: Quinapril
Drug: Placebo — Placebo will be given in a capsule form once daily for 16 weeks.
  Arms: Placebo

SUMMARY:
INDICATION Microvascular angina. OBJECTIVES To investigate the effect of ACE (angiotensin converting enzyme) inhibition (quinapril) in improving coronary microvascular function.

PATIENT POPULATION Women who meet the National Heart, Lung and Blood Institute-sponsored WISE (Women Ischemia Syndrome Evaluation) study criteria of chest discomfort, coronary flow reserve limitations and evidence for myocardial ischemia in the absence of significant coronary artery stenosis.

STUDY DESIGN A prospective, randomized, placebo-controlled, comparative trial. TREATMENT Quinapril 80 mg/d versus placebo for four months. PRIMARY EFFICACY PARAMETER(S) Coronary flow reserve (CFR) at Week 16 adjusted for baseline CFR, treatment group assignment, site-specific variables, and site by treatment effects.

SECONDARY EFFICACY PARAMETERS Week 16 change in chest discomfort as measured by the Seattle Angina Questionnaire adjusting for baseline values, site, and site by treatment effects.

SAFETY PARAMETERS Hematology, blood chemistries, blood pressure and pulse, and frequency and occurrence of adverse events.

STATISTICAL RATIONALE AND ANALYSIS A statistical rationale for the number of patients in the study has been provided. Interim analyses are planned after 15 patients have been enrolled in each group.

ANTICIPATED TOTAL NUMBER OF PATIENTS 78 (39 per group). ANTICIPATED NUMBER OF PATIENTS AT EACH SITE Approximately 26

DETAILED DESCRIPTION:
A prospective, randomized, placebo-controlled, comparative trial evaluating the effects of ACE inhibition on microvascular function in women with coronary flow reserve limitations and chest discomfort. Women who are enrolled in the WISE study can be enrolled into this ancillary study if they meet the study criteria. Women not enrolled in the WISE study can also be entered into this ancillary study as long as they too meet the study criteria. After WISE evaluations including symptom assessment using the Seattle Angina Questionnaire (SAQ) and documented reduced coronary blood flow reserve (<3.0 velocity), patients will be randomized to double-blind placebo or quinapril (started at 40 mg/d and titrated to 80 mg/d by the end of the first week). After treatment on the maximum tolerated dose for 16 weeks, patients will be reevaluated with coronary angiogram with coronary flow reserve measurements and assessment of angina using the SAQ.

ELIGIBILITY:
Inclusion Criteria:

1. Non pregnant women with chest discomfort 21 to 75 years of age from diverse racial/ethnic groups.
2. Suspected ischemic heart disease (IHD) but no severe coronary stenosis (> 50% diameter reduction) on coronary angiography used to qualify for WISE.
3. Coronary flow reserve limitation (<3.0 velocity).

Exclusion Criteria:

1. Women who are breast-feeding or who are pregnant. Women of childbearing potential may be enrolled but must agree not to become pregnant during the course of the study and must practice a method of birth control considered reliable by the investigator. If established on hormonal contraceptives for more than 3 months, patients will be allowed to participate providing this therapy remains constant throughout the study. If a patient becomes pregnant or begins breast-feeding during the study, she must be withdrawn immediately.
2. Acute ischemic syndrome defined as acute myocardial infarction (MI) (by enzyme or electrocardiogram (ECG) criteria) or unstable angina within 1 month of entry.
3. Uncontrolled moderate hypertension: Sitting blood pressure >160/95mmHg with measurements recorded on at least 2 occasions (for blood pressure control, patients must first be stabilized, preferably with a diuretic, and kept on that dosing regimen throughout participation in the study).
4. Severe heart failure defined as New York Heart Association (NYHA) Class III or IV on treatment.
5. Coronary revascularization by either coronary artery bypass grafting (CABG) or percutaneous transluminal coronary angioplasty (PTCA) or Stent Placement.
6. Conditions likely to influence outcomes independent of IHD: Severe lung, renal (creatinine >3.0) or hepatic disease, surgically uncorrected significant congenital or valvular heart disease and other disease likely to be fatal or require frequent hospitalization within the next six months.
7. Adherence or retention reasons: Recent alcoholism or drug abuse, psychiatric illness including severe depression, dementia, active participation in any other research trial other than WISE, unwilling to complete follow-up evaluation including repeat testing.
8. Hypersensitivity to any medications to be used in the study (e.g. angioedema to ACE-I).
9. Documented obstructive hypertrophic cardiomyopathy.
10. Aortic stenosis (valve area <1.5cm).
11. LV dysfunction (ejection fraction <=35%).
12. History of cocaine or amphetamine abuse.
13. ACE-I or angiotension 1 (AT-1) receptor blocker use within 30 days or need for continued ACEI/AT-1RB use.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2000-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Adjusted coronary flow reserve at Week 16

SECONDARY OUTCOMES:
Chest pain as measured by a Seattle Angina Questionnaire adjusted for baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Pauly DF, Johnson BD, Anderson RD, Handberg EM, Smith KM, Cooper-DeHoff RM, Sopko G, Sharaf BM, Kelsey SF, Merz CN, Pepine CJ. In women with symptoms of cardiac ischemia, nonobstructive coronary arteries, and microvascular dysfunction, angiotensin-converting enzyme inhibition is associated with improved microvascular function: A double-blind randomized study from the National Heart, Lung and Blood Institute Women's Ischemia Syndrome Evaluation (WISE). Am Heart J. 2011 Oct;162(4):678-84. doi: 10.1016/j.ahj.2011.07.011. Epub 2011 Sep 6. PMID 21982660